

## Statistical analysis

IBM SPSS version 23 will be used for the statistical analysis. The sociodemographic and clinical characteristics of the patients will be analyzed using descriptive statistics. Differences between the two intervention groups (IPT+EMT versus TAU) will be analyzed using the  $X^2$  test (or Fisher's test where n < 5) for categorical variables and the Student's t test or Mann-Whitney t0 test (depending on the distribution of the data) for continuous variables.

Effect sizes will be calculated for differences in both conditions of treatment based on Cohen's d or r [36] for Student's t test and the Mann-Whitney U test, respectively. The results will be interpreted as small if d values are between .20 and .49 and if r values are 0.10-0.29, medium if d values are between .50 and .79 and if r values are 0.30-0.49, and large if d values are higher than .80 and if r values are >0.50

The maintenance of the results in the experimental group in the 6- and 12-month follow-up will be analyzed with repeated measures t-test paired sampled statistic or Wilcoxon signed-rank test depending on the distribution of the data.